CLINICAL TRIAL: NCT00219102
Title: A 12-week, Randomized, Double-blind, Placebo Controlled, Parallel Group Study Evaluating the Efficacy & Safety of Aliskiren in Patients With Diabetes & Hypertension Not Adequately Responsive to the Combination of Valsartan 160 mg & Hydrochlorothiazide 25 mg
Brief Title: A Clinical Study to Evaluate Safety & Efficacy of the Combination of Aliskiren, Valsartan & Hydrochlorothiazide in Diabetic Hypertensive Nonresponder Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2310
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2011-02

CONDITIONS: Hypertension; Diabetes
Keywords: Hypertension,; diabetes,; aliskiren,; blood pressure,; valsartan,; hydrochlorothiazide
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To evaluate the blood pressure lowering effect and safety of aliskiren used in combination with valsartan/hydrochlorothiazide in diabetic patients with essential hypertension, not adequately responsive to the combination of valsartan and hydrochlorothiazide

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients with a documented diagnosis of Type 1 or Type 2 diabetes mellitus.
* Patients who are eligible and able to participate in the study

Exclusion Criteria

* Severe hypertension
* Uncontrolled diabetes type I and II
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident.

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336
Dates: Start 2005-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 12 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 12 weeks
Change from baseline in systolic and diastolic blood pressure after 6 weeks
Diastolic blood pressure of < 80 mmHg or a reduction from baseline of diastolic blood pressure of > 10 mmHg after 12 weeks
Achieve mean sitting blood pressure control target of < 130/80 mmHg after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Investigative Site, Salisbury, North Carolina, United States
- Investigative Site, Kortrijk, Belgium
- Investigative Site, Bucharest, Romania
- Investigative Site, Madrid, Spain
- Investigative Site, Stockholm, Sweden
- Novartis Pharmaceuticals, Basel, Switzerland
- Investigative Site, Kiev, Ukraine

REFERENCES:
- [Derived] Drummond W, Sirenko YM, Ramos E, Baek I, Keefe DL. Aliskiren as add-on therapy in the treatment of hypertensive diabetic patients inadequately controlled with valsartan/HCT combination: a placebo-controlled study. Am J Cardiovasc Drugs. 2011 Oct 1;11(5):327-33. doi: 10.2165/11591970-000000000-00000. PMID 21846154